CLINICAL TRIAL: NCT07193355
Title: Effects of Motor Imagery Training on Kinesiophobia, Gait, and Balance in Parkinson's Disease Patients
Brief Title: Effects of Motor Imagery Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, Associate Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Parkinson lower extremity
Record Dates: First submitted 2025-09-12; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-07

CONDITIONS: PARKINSON DISEASE (Disorder); Mental Imagery; Gait Balance
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): 'Mental Imagery Application Protocol' will be applied to this group. The timed up and go test (TUG) and gyko test will be used as mental chronometry tests with the patients of parkinson diesase.Therefore, the walking mental imagery protocol will be applied to this group.
  Interventions: Other: Mental Imagery Application Protocol
- control group (No Intervention): This group will have routin medical treatment.

INTERVENTIONS:
Other: Mental Imagery Application Protocol — Before the GYKO test, the patient will be asked to perform mental imagery to visualize a 3-meter distance for five cycles, and the time will be recorded. The TKYT will be administered according to standard protocols.
  Mental Imagery Application Protocol:
  1. Awareness:
     The therapist will show a video of a typical normal gait for an adult male or female without pathology and compare it with a video of the patient's own gait.
  2. Problem Identification/Explanation In the EG, subjects will identify gait problems and compare their gait with their typical gait. They will then use the comparative information for feedback.
  3. Progressive Relaxation
  4. Mental Imagery of Gait
  5. Physıcal Performance Of The gait This protocol will be implemented the day after the initial assessment and will be conducted in 12 training sessions of no more than 90 minutes, three times per week for 4 weeks.
  Arms: study group

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disease, characterized pathologically by the progressive loss of dopaminergic neurons in the substantia nigra and clinically by the presence of motor symptoms such as bradykinesia, resting tremor, and/or rigidity. Among the motor deficits frequently observed in PD, patients are known to frequently report difficulties with manual dexterity.Typical features of balance deficits in PD include decreased sway, decreased base of support, rigidity, abnormal intersegmental coordination, and postural misalignment. Related somatosensory deficits in PD include problems orienting to and processing sensory and somatosensory information.Motor imagery (MI) is the imaginal execution of motor activities or the activation of specific muscles in the absence of any explicit feedback. This area of rehabilitation has been shown to be effective in improving and developing motor skills in many neurological conditions where patients exhibit motor recognition and execution impairments. MI can be applied at all stages of recovery from PD, is highly effective in movement-related pathologies, and can be performed independently.Studies evaluating the effect of mental imagery training on balance measures in PD are limited. One study evaluating the effect of combined MI-physical therapy versus physical therapy alone group treatment noted positive trends toward balance improvements in the combined group. In a case study of a single participant with PD, a 3-month neurocognitive rehabilitation program incorporating mental imagery over 20 sessions resulted in balance improvements and a reduced risk of falls in both the "OFF" and "ON" phases, as measured by the Tinetti Balance and Gait Assessment Scale.The aim of this study is to investigate the effects of motor imagery training on kinesiophobia, walking and balance in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 40-75 diagnosed with idiopathic PD, with a Modified Hoehn & Yahr (m-HY) scale stage ≤4, and a score of ≥22 on the Mini Mental State Examination for those with formal training and ≥18 for those without formal training;
* Individuals with no other known neurological and/or systemic disease;
* Individuals without any upper extremity contractures;

Exclusion Criteria:

* Individuals with diagnosed and/or treated psychiatric illnesses;
* Individuals who are taking neuroleptic medications or antidepressants;
* Individuals with orthopedic conditions such as severe dyskinesia, carpal tunnel syndrome, tendon injuries, and finger amputations that interfere with manual dexterity tests; rheumatological conditions such as rheumatoid arthritis and osteoarthritis; and individuals with any neurological disease other than PD.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Mental Chronometry with Timed up Go Test and Gyko device | first day of the assessment and after the end of the treatment protocol (in the 5th week of the assessment) .
  Mental chronometry is a method considered more objective than questionnaires in the assessment of MI, measuring imagery time. In other words, it examines the time difference between the actual physical execution of a movement and the mental imagery of the same movement. In the calculated mental chronometry value, a value of zero indicates perfect synchrony between motor imagery and motor execution. Values above zero indicate that the task was performed faster during motor imagery than during motor execution, and values below zero indicate that the task was performed slower during motor imagery than during motor execution. Patients' actual walking times (MIT) and imagery times (MET) are recorded. The difference in time and the mental chronometry ratio are calculated, and the mental chronometry ratio is evaluated using the following formula.In our study, the timed up and go test (TUG) and the gyko test will be used as mental chronometry tests.
Tampa Kinesiophobia Scale | first day of the assesment and the 5th week of the treatment protocol.
  The Tampa Kinesiophobia Scale (TKS) is a 17-question checklist developed to measure fear of movement and re-injury. Items are scored on a 4-point Likert scale (1: Strongly disagree, 4: Strongly agree). A total score is calculated by reversing items 4, 8, 12, and 16. A person receives a total score between 17 and 68. A total score of 37 points or higher indicates a high level of kinesiophobia. As a participant's score increases, so does the severity of their kinesiophobia. The use of the total score is recommended in studies. A Turkish version of the scale was developed and its reliability study was conducted in 2011.
The Gyko Device | baseline and the 5th week of the treatment protocol.
  This device, manufactured by Mikrogate and manufactured in Italy, is used as a portable inertial measurement unit for motion analysis and postural stability assessment. The displacement of the center of gravity is analyzed using a computer using a sensor placed on a sling. The patient is asked to walk for 30 seconds.

SECONDARY OUTCOMES:
The Kinesthetic and Visual Imagery Questionnaire (KVIQ)-short form | first day of the assesment and 5th week of the treatment protocol.
  The Kinesthetic and Visual Imagery Questionnaire (KVIQ), Short Form, was developed to determine the extent to which individuals visualize and feel the imaged movements. It consists of a total of 10 movements measuring five visual and five kinesthetic imagery skills (24). The questionnaire is not a self-report measure but is administered by an assessor. All movements were assessed in a sitting position. The assessor first performed the relevant movement on themselves and then asked the participant to perform the same movement only once. The participant then visualized the movement and rated the visual clarity or intensity of sensations on a five-point ordinal scale. Higher scores indicate greater visual clarity or intensity of sensations.
Modified Hoehn & Yahr (m-HY) Scale | first day of the assesment and the 5th week of the treatment protocol.
  PD disability will be assessed with the m-HY scale: stage 1.0 (unilateral involvement only); stage 1.5 (unilateral and axial involvement); stage 2.0 (bilateral involvement without balance impairment); stage 2.5 (mild bilateral disease with improvement on pull test); stage 3.0 (mild to moderate bilateral disease; some postural impairment; physically independent); stage 4.0 (severe disability; still able to walk or stand unaided). Symptom severity in PD was graded using the Unified Parkinson's Disease Rating Scale (UPDRS): part I (mental dysfunction and mood); part II (activities of daily living); part III (motor component); part IV (treatment-related complications)
sosyodemographic form | first day of the assesment and the 5th week of the treatment protocol.
  Medical history (disease duration and symptoms), demographic information will be recorded.
Unified Parkinson's Disease Rating Scale (UPDRS) | first day of the assesment and the 5th week of the treatment protocol.
  Symptom severity in PD is rated using the Unified Parkinson's Disease Rating Scale (UPDRS). Several items on this scale assess upper extremity and hand function. The Activities of Daily Living section assesses handwriting, cutting food, and grasping utensils. The Motor section assesses finger tapping, hand movements, and rapid alternating hand movements. These test items are scored from 0 to 4, with 4 representing maximum impairment and 0 representing normal movement ability. The UPDRS is comprised of subsections: Section I (mental dysfunction and mood); Section II (activities of daily living); Section III (motor); and Section IV (treatment-related complications).
Mini Mental State Examination (MMSE) | first day of the assesment and the 5th week of the treatment protocol.
  This test was developed by Folstein in 1975. Its Turkish validity and reliability study was conducted by Güngen et al. in 2002. The Mini Mental State Examination (MMSE), which is quite suitable for screening cognitive function in the elderly and assesses cognitive functions in five separate areas (orientation, registration, attention and calculation, recall, and language), is frequently used. A score below 24 on the MMSE indicates dementia, 24-26 indicates mild cognitive impairment, and 26 or above indicates normal cognitive function.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Sütçü imam University, Kahramanmaraş, Onikişubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No